CLINICAL TRIAL: NCT02598518
Title: Integrating Combined Therapies for Persons With Co-occurring Disorders
Acronym: ICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mark McGovern, Study Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AA023001-01A1 (NIH); 1R21AA023001-01A1 (NIH)
Record Dates: First submitted 2015-10-27; First posted 2015-11-06 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Alcohol Use Disorder; Mental Health Disorder
Keywords: Integrating Combined Therapies; Alcohol Use Disorder; Mental Health Disorder
MeSH Terms: conditions — Alcoholism; Mental Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrating Combined Therapies (Experimental): Integrating Combined Therapies (ICT) is a 10-session, manual-guided individual therapy. ICT has three phases designed to address substance use, psychiatric problems and their interactions. MET is the first phase (2 sessions) and is focused on assessment, feedback and securing motivation to address problems and take steps. CBT is the second phase (5 sessions) and incorporates patient education and functional analysis, develops coping skills, teaches methods to challenge beliefs, and activates alternative behaviors. TSF (3 sessions) is focused on maintaining recovery and engaging in community-based recovery activities. Although ICT has core components, its application is flexible to accommodate the unique needs and problems of individual patients (and their comorbidities).
  Interventions: Behavioral: Integrating Combined Therapies
- Standard Care (Active Comparator): Standard Care (SC) is the typical outpatient treatment that the patient would receive ordinarily at the identified addiction treatment program. SC service operates using the American Society of Addiction Medicine criteria (9 hours per week); group and individual sessions focused on motivation to address substance use, education about the consequences of substance use on major life areas, education about the disease concept and brain changes associated with addiction, exposure to information about social and family relationships and recovery, and relapse prevention skills.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Integrating Combined Therapies — Individual Integrating Combined Therapies, approximately 10 sessions, one session per week
  Other Names: ICT
  Arms: Integrating Combined Therapies
Behavioral: Standard Care — Standard Care, individual or group therapy, approximately 9 hours per week for 3 months.
  Other Names: SC
  Arms: Standard Care

SUMMARY:
The purpose of this study is to assess the effectiveness and implementability of ICT for co-occurring alcohol use and mental health disorders within community addiction treatment, as delivered by routine community addiction clinicians.

DETAILED DESCRIPTION:
The proposed study will evaluate the effectiveness and implementability of a manual-guided integrated psychosocial treatment, Integrating Combined Therapies (ICT). ICT is an adaptation of the Combined Behavioral Intervention (CBI) from NIAAA Project COMBINE, and expands CBI's indication for alcohol problems to extend to drug use and the most common psychiatric problems in addiction treatment. ICT is designed to be transferable to routine care settings and for delivery by the existing workforce. Findings from a 2014 study provide a signal for ICT effectiveness and implementation.

We intend to randomly assign 76 eligible patients in outpatient addiction treatment to ICT adapted standard care (ICT+SC) versus standard care only (SC). There are 2 specific aims for this study:

Aim 1: Relative to standard care alone, to evaluate if patients receiving ICT have more significant reductions in alcohol use and severity as measured by the 90-day Timeline Follow Back (TLFB), Addiction Severity Index (ASI), and Short Inventory of Problems (SIP).

Aim 2: Relative to standard care alone, to evaluate if patients receiving ICT have more significant reductions in psychiatric symptom severity, as measured by the Brief Symptom Inventory (BSI) adn the ASI psychiatric severity composite.

This study involves a two-group repeated measure design. This study is a randomized controlled trial. The investigators plan to examine the outcomes associated with ICT versus standard care among patients receiving outpatient addiction treatment services. The investigators will employ assessments at baseline, four-month follow-up, and seven-month follow-up. Eligible participants will be randomly assigned to ICT therapy (plus standard care) or standard care, and all will be followed for the research assessments regardless of whether they drop out of treatment early (whenever possible).

Patients admitted to the participating addiction treatment program are routinely screened for an alcohol use disorder using the AUDIT and a mental health disorder using the MMS. These forms are collected by clinic staff and scored for alcohol use disorder (AUDIT: 8 or greater) and mental health disorder (MMS: 6 or greater). Patients meeting the threshold criteria on the AUDIT and MMS measures are approached by clinic staff about potential interest in the study. If they wish to learn more about the study, the research assistant is contacted, a suitable time is arranged, and the patient engaged in the process of informed consent.

If consent is granted, the participant completes the baseline assessment. The baseline assessment consists of measures gathered via interview by a member of the research team, self-administered surveys completed directly by the participant, and review of the participant's medical record to extract substance use, treatment history, and chart diagnoses.

The interview portion of the assessment consists of :

* Standardized interview designed to assess mental health diagnoses: Structured Clinical Interview for DSM5 (SCID).
* A urine screen and breathalyzer to test for alcohol and other drugs.
* Standardized follow-back method for gathering data on recent alcohol and drug use: Timeline Follow-back calendar (TLFB)

The self-administered portion of the assessment consists of measures designed to assess:

* Alcohol and drug use, as well as associated problems in other life areas such as medical, employment, legal, social, and psychiatric: Addiction Severity Index
* Psychiatric symptoms: Brief Symptom Inventory (BSI)
* Mental health disorders: Modified MINI Screen (MMS)
* Negative consequences of alcohol and substance use: Short Inventory of Problems- Alcohol and Drugs (SIP-AD)
* Substance use symptoms and problems: Brief Addiction Monitor (BAM)
* Treatment utilization: Recent Treatment Survey (RTS)

If the participant continues to meet criteria for a mental health disorder (i.e. SCID interview confirms diagnosis of DSM5 mental health disorder, he or she is randomized to receive the study ICT therapy or standard care (SC)

Research assessments are then also conducted at four months and seven months post baseline assessment. The follow-up assessments will consist of the same measures administered at baseline, with the exception of the SCID interview.

The investigators plan to randomize approximately 76 participants in the study.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old;
2. Evaluated and admitted to outpatient addiction treatment services at RMHS Evergreen program and meets criteria for any alcohol or substance use disorder;
3. Screened positive for an alcohol problem on the Alcohol Use Disorders Identification Test (AUDIT) (score of 8 or higher) (screening instrument);
4. Screened positive for a mental health problem on the Modified MINI Screen (MMS) (score of 6 or higher) (screening instrument);
5. Diagnoses confirmed by SCID (diagnostic interview); AND
6. Willing and able to provide informed consent.

Exclusion Criteria:

1. They have acute psychotic symptoms and are not appropriately connected with mental health services;
2. They have had a psychiatric hospitalization or suicide attempt within the past month (however, if the hospitalization or attempt was directly related to substance intoxication or detoxification and the person is currently stable, they are eligible); OR
3. They have unstable medical or legal situations that would make participation for the full duration of the study highly unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Decrease from baseline in alcohol use (90-day Timeline Follow Back (TLFB) at 4-months and at 7-months | Baseline, 4-month, 7-month follow-up
Decrease from baseline in alcohol use severity (ASI; alcohol severity composite) at 4-months and at 7-months | Baseline, 4-month, 7-month follow-up
Decrease from baseline in alcohol use severity (Short Inventory of Problems (SIP)) at 4-months and at 7-months | Baseline, 4-month, 7-month follow-up
Decrease from baseline in psychiatric symptom severity (ASI; Psychiatric Severity Composite) at 4-months and at 7-months | Baseline, 4-month, 7-month follow-up
Decrease in psychiatric symptom severity (Brief Symptom Inventory (BSI)) at 4-months and 7-months | Baseline, 4-month, 7-month follow-up

SECONDARY OUTCOMES:
Decrease from baseline in drug use (90-day TLFB) at 4-months and at 7-months | Baseline, 4-month, 7-month follow-up
Decrease from baseline in positive toxicology screen (urine drug screen) at 4-months and at 7-months | Baseline, 4-month, 7-month follow-up
Decrease from baseline in drug use severity (ASI; Drug Severity Composite) at 4-months and 7-months | Baseline, 4-month, 7-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mark P. McGovern, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Evergreen - Rutland Mental Health, Rutland, Vermont, United States